CLINICAL TRIAL: NCT05723289
Title: Evaluation of the Feasibility of Remote Monitoring of Cough Assist Devices in Paralytic and Neuromuscular Patients Treated at Home
Brief Title: Evaluation of the Feasibility of Remote Monitoring of Mechanical In-exsufflation Devices in Paralytic and Neuromuscular Patients Treated at Home.
Acronym: TELE-INEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KerNel Biomedical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A01442-41
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Neuromuscular Diseases; Scoliosis
Keywords: Neuromuscular; scoliosis
MeSH Terms: conditions — Neuromuscular Diseases; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MI-E Telemonitoring — Daily telemonitoring using a ad-hoc communicating device

SUMMARY:
The implementation of an mechanical in-exsufflator device (MI-E) requires specific expertise because it is a complex device that requires fine-tuning of the settings according to different clinical situations to optimize its effectiveness. Generally, it is performed by experienced physiotherapists in neuromuscular disease reference centers or directly at home via medical-technical home care providers.

Treatment data is recorded by the machine at each MI-E session, which may be daily or less frequent, depending on the patient's dependency. All of this information can be accessed by manually downloading the data from the SD card that comes with each MI-E machine. Therefore, the retrieval of this information systematically requires the visit of staff to the patient's home.

To date, compliance with these devices is not regularly measured since there is no means of telecommunication allowing remote monitoring of these therapies, whereas technological development in the field of remote monitoring has allowed remote monitoring of patients with sleep apnea syndrome treated with continuous positive airway pressure (CPAP) and, more recently, of some patients with chronic respiratory insufficiency treated with invasive ventilation (NIV). These developments are transforming on the one hand the follow-up of patients under NIV at home by the medical and paramedical teams and on the other hand the financial coverage by the health insurance organizations (ETAPES programs). Within the framework of NIV therapy, we think that remote monitoring of the quality of the sessions, i.e. measurement of peak expiratory flow, insufflated volumes, frequency and duration of the sessions, could facilitate and improve the follow-up of these patients for the medical-technical providers, the expert physiotherapists and the doctors of the reference centers. It is still too early to assume the extent to which data from remote monitoring of MI-E devices would improve patient follow-up. Nevertheless, given the increasing number of devices installed over the past several years, it is likely that the issue of telemonitoring will become a central issue. Thus, in this observational trial, we propose to evaluate the feasibility of a simple system of remote monitoring of MI-E devices in non-therapy-naive patients, with the objective of assessing the barriers and limitations of remote monitoring in this population.

Primary aim is to evaluate the feasibility of remote monitoring of data from the MI-E device used in the patient's home in neuromuscular diseases.

Patients will be identified by the investigators using the AGIR à dom software package (medical-technical follow-up file). If the patient accepts, the information and no-objection form will be sent to them electronically or by mail following this call, and at least 3 days before their scheduled appointment.

During the patient's usual follow-up visit, if the patient does not object to participating in the study, AGIR staff in dom will install the device. This visit will take place in the patient's home. During this visit, a SanDisk (SD) Eye-Fi SDHC 4GB + WiFi Class4 memory card will be inserted into the port provided, in place of the memory card already present in the MI-E device. Then a Raspberry Pi 4 Model B will be placed in the room where the MI-E device is normally used by the patient, and connected to a power source (accessible electrical outlet in the room). The wifi SD card, which uses the device's power supply, will communicate with the Raspberry Pi via the wifi network and upload the recorded data each time the MI-E device is used.

After 90 days, a routine recovery visit will be scheduled. AGIR à dom staff will replace the wifi SD card installed during the D0 visit with the standard SD card originally provided with the MI-E device. The data locally on the SD Wifi card will then be downloaded for analysis and comparison with the data being uploaded

DETAILED DESCRIPTION:
Perspectives

Democratizing remote monitoring of cough devices would:

Potentially decrease the costs associated with data retrieval Encourage the establishment of centers of expertise where expert practitioners could follow multiple patients (e.g., at the provider's site).

To study the relationship between certain data from the MI-E (use, adjustment of settings, peak expiratory flow or insufflated volume).

The development of an automated analysis system for predictive data (increase in bronchial congestion, inefficiency of the device) to optimize the follow-up of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient over 18 years of age
* Patients with neuromuscular or paralytic disease
* Patient previously treated with an E70 in-exsufflation device (Philips Respironics)
* Patient with known use of the E70 in-exsufflation device at least once a week, excluding episodes of infection.
* Patient followed by AGIR at home
* Patient willing to participate in the research after adequate information and delivery of the information note.
* Patient affiliated to the social security system or beneficiary of such a system.

Exclusion Criteria:

* No internet solution at home (adsl/fibre box)
* Technical inability to connect the computer to the Internet by Ethernet cable
* Person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure (patient under guardianship or curatorship) Article L1121-8.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuromuscular disease or paralytic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of remote monitoring of data from the MI-E device used in the patient's home. | 90 days
  The difference between the number of sessions of device use uploaded and the actual number of sessions performed, collected from the internal memory of the device.

SECONDARY OUTCOMES:
Compare cost of telemonitoring versus cost of monitoring by a technician in the patient's home | 90 days
  Cost of telemonitoring equipment, time required for installation or troubleshooting compared to the cost of usual monitoring requiring home visit(s)
Describe the type of data collected through remote monitoring of MI-E devices | 90 days
  Daily or weekly usage times (minutes), detailed cough expiratory flow data (l/min) and detailed inspiratory volume data (liters)
Identify the factors limiting the implementation of telemonitoring | 90 days
  Proportion of non-communicating devices, proportion of disconnections or lack of data feedback

CONTACTS AND LOCATIONS:
Locations (1):
- Borel Jean-Christian, Meylan, France